CLINICAL TRIAL: NCT06582498
Title: Life S-Can: a Novel Clinical Tool to Effectively Assess Individual Needs in Cancer Survivorship Care and Improve Quality of Life in Cancer Survivors
Brief Title: Short Questionnaire to Assess Individual Needs in Cancer Survivors in a Clinical Setting
Acronym: LIFE S-CAN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Alice Mary Lillian Chaplin, Principal Investigator, Fundació d'investigació Sanitària de les Illes Balears
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMP23/01
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cancer Survivors
Keywords: Cancer survivorship; Screener; Diet; Physical activity; Psychosocial distress
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A random allocation system will be applied to participants, which will be allocated to the Low Intensity Intervention Group (LIIG) or the Active Intervention Group (AIG). Both groups will attend a first, baseline visit offered to all participants with a trained dietitian, who will administer the Life S-Can questionnaire and a series of validated questionnaires. The LIIG will receive the standard care and recommendations already provided by the Oncology Department of the hospital and a set of recommendations for cancer prevention offered by the WCRF, the AICR and the ACS. The AIG will receive the same recommendations as the LIIG and will be offered to see an oncological dietitian (diet domain), a physical activity health professional (physical activity) and/or a psychologist (psychosocial distress) for two visits (one individual, one group session). All participants will attend a final visit after 3 months to collect data on feasibility, acceptability and efficacy of the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Consists of participants (50% of the total recruited) which will receive the Active Intervention.
  Interventions: Behavioral: Active intervention
- Low-intensity intervention (Active Comparator): Consists of participants (50% of the total recruited) which will receive the Low Intensity Intervention.
  Interventions: Behavioral: Low-intensity intervention

INTERVENTIONS:
Behavioral: Active intervention — This group will receive a pamphlet with diet and lifestyle recommendations for cancer survivors at randomization (2nd visit). Furthermore, they will be offered 3 individual sessions with health professionals (oncological dietitian, sports therapist, and oncological psychologist) and 3 group sessions with the same professionals. The duration of the individual visits is expected to be 45-60 minutes approximately, and group sessions will be planned for 1.5h duration approximately.
  Arms: Active intervention
Behavioral: Low-intensity intervention — This group will receive a pamphlet with diet and lifestyle recommendations for cancer survivor at randomization (2nd visit). These recommendations are all based on information from the World Cancer Research Fund, the American Institute for Cancer Research, and the American Cancer Society.
  Arms: Low-intensity intervention

SUMMARY:
The rate of cancer survivorship is increasing, posing the need to create high quality survivorship care plans. Traditionally, follow-up of cancer survivors has focused on detection of cancer recurrence or new cancers, but often it does not fully address behavioural and psychosocial elements which could improve quality of life (QoL) and potentially decrease recurrence risk. There is a current lack of short, validated screeners to assess diet, lifestyle and other behaviours that might influence QoL and prognosis in cancer survivors. The hypothesis of this project is that the creation of a screener with the capacity to rapidly, validly and effectively assess nutritional factors, lifestyle, sleep quality and psychosocial distress in cancer survivors could be useful to identify individuals who may need further care and support. The aim is to create a valid and rapid tool (Life S-Can) to evaluate a total of seven domains (body composition, physical activity, diet, alcohol intake, smoking, sleeping behaviour and psychosocial distress) in cancer survivors for its use in a clinical setting to improve survivorship care and QoL. The project is divided into three phases and will be carried out in one year at the University Hospital Son Espases (HUSE) (Palma, Spain). The objective of Phase I is to design the screener, which will be administered to a small convenience sample to determine comprehension, clarity and usefulness. In Phase II, Life S-Can will be validated in cancer survivors (n=100) at HUSE and a pilot intervention will be carried out with the objective to test the feasibility of a larger intervention to effectively implement Life S-Can in clinical settings to improve QoL in cancer survivors. For this, patients will be recruited by the Oncology Department and will be invited to attend the Clinical Trials Unit for an exhaustive assessment. A research dietitian will administer Life S-Can and will then collect data using validated questionnaires and objective measurements to compare to the data obtained with the Life S-Can screener. Participants will then be randomly allocated to either the Low Intensity Intervention Group (LIIG) or Active Intervention Group (AIG). LIIG patients will receive standard care and advice given to cancer survivors, and AIG patients will receive personalised feedback (by means of individual and group sessions) in order to improve their body composition, physical activity, diet, alcohol intake, and psychosocial elements based on their answers, by trained professionals. Patients of both groups will also answer both Life S-Can and validated questionnaires at baseline and after three months. Outcome measurements will be indicators of feasibility (completion of questionnaires), acceptability (by patients, health professionals), behavioural changes (diet, physical activity, psychosocial distress) and QoL. Finally, Phase III consists of a qualitative study conducted in cancer patients and health professionals to obtain data to design an implementation study. Cancer survivors care should be multifactorial; however, often, due to time constraints and clinical burden, health professionals might not assess certain aspects relevant for cancer survivors' QoL, such as nutritional status, diet, physical and mental health adequately. Life S-Can will enable clinicians, health practitioners, charities and other stakeholders work with cancer survivors early-on and refer them to adequate health and mental care teams and resources.

DETAILED DESCRIPTION:
The aim of this project is to develop a valid and rapid screening tool (Life S-Can) with the capacity to evaluate a total of seven domains (body composition, physical activity, diet, alcohol intake, smoking, sleeping behaviour and psychosocial distress) in cancer survivors for its use in a clinical setting to improve survivorship care and QoL. The project is divided into four specific aims (SA) and will be carried out in one year at the University Hospital Son Espases (HUSE) (Palma, Spain).

SA1: Develop a short screener (Life S-Can) to evaluate body composition, physical activity, diet, alcohol intake, smoking habits, sleeping behaviour and psychosocial distress in cancer survivors.

SA2. Determine relative and construct validity of individual domains and total score of the Life S-Can in cancer survivors using data obtained from validated and objective measurements.

SA3. Carry out a pilot intervention study in cancer survivors to determine the feasibility, acceptability and efficacy of Life S-Can.

SA4. Carry out a qualitative study in cancer survivors and health professionals to design an implementation study.

The project herein presented proposes three phases: tool development (Phase I); validation of the tool (Phase II - validation and pilot intervention study); and qualitative (Phase III).

PHASE I: Phase I refers to SA1.

Recruit an expert panel: Together with the Principal Investigator, five key personnel have been listed in this project, all of whom carry out research at the Health Research Institute of the Balearic Islands (IdISBa, Spain) together with other duties (university professor, medical doctor). Key personnel not contemplated as researchers in this project include international experts in nutrition and cancer and will be consulted throughout the project. Cancer survivors will also be contacted at this stage (through the hospital) to involve them in the design stage.

Elements of the intervention at discussion: A series of meetings, semi-structured interviews and panel groups will be planned with expert panel members and non-scientific actors to define the best intervention. Elements to be defined during this stage are: scoring of the individual domains of Life S-Can herein studied and traffic-light system (good, intermediate and non-adherence, which will direct the intervention and health professionals to be visited), monitoring of patients, pipeline, feedback, appointment system, Clinical Trials Unit and data collection.

PHASE II:

Phase II consists of two objectives: a validation study (SA2) and a pilot intervention study (SA3). The validation study will consist of three visits to the research/hospital facility. The first visit will be at the Clinical Trials Unit, will take approximately 1 h and will be divided into three parts: 1) Administration of Life S-Can; 2) Administration of validated questionnaires; and 3) Obtain objective measurements of the patient. The second visit will also be at the Clinical Trials Unit and will take approximately 10-15 minutes. Participants will be asked to return the accelerometer and complete the Life S-Can questionnaire again (reproducibility). At this visit, patients will be randomly allocated to the Low Intensity Intervention Group (LIIG) or Active Intervention Group (AIG). The third and final visit will also be at the Clinical Trials Unit and will take approximately 30 minutes. The participant will be asked to answer the Life S-Can again, together with other questionnaires (QLQ-C30) and anthropometric measurements, to measure changes in QoL.

The pilot intervention study (SA3) will be designed using a multi-disciplinary approach, whereby knowledge and expertise in oncology, nutrition, epidemiology, psychology and psychometry, validation and implementation will be called upon. In addition, the views and experiences of cancer patients and patient organizations are essential in designing an effective intervention; hence non-scientific authors will be contacted and included in this phase.

This intervention phase is divided into three stages: intervention design, patient recruitment and group allocation and intervention. Participation in this study will entail visits to the Clinical Trials Unit at IdISBa, located within the Hospital Universitari Son Espases. When possible, visits will be coordinated with other routine appointments at the hospital in order to reduce as much as possible the burden on the participant. Dietary, physical activity and psychologic interventions will be carried out by in-house researchers (trained oncological dietitian) and external health professionals.

Participants allocated to the LIIG will receive routine advice offered by their oncological care team and a set of standard recommendations offered by the World Cancer Research Fund, the American Institute for Cancer Research and the American Cancer Society. Participants in the AIG will also receive this, and will also be offered the chance to visit an oncological dietitian, a physical activity health professional and a psychologist (one individual session, and one group session).

At the final visit, Life S-Can and QLQ-C30 questionnaires will be administered again in order to determine any changes or impact on lifestyle and quality of life. Information regarding feasibility and acceptability of the intervention will be collected from participants.

PHASE III. The aim of the qualitative study is to design an implementation study.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old; men & women; able to read and understand Spanish; prior diagnosis of cancer (stages I to III); have completed all systemic treatment (surgery, chemotherapy, radiation therapy) at least ≥3 months prior to the study start date; be currently considered cancer free; able to attend visits at HUSE.

Exclusion Criteria:

* Ongoing cancer or cancer treatment; have a debilitating medical or psychiatric illness; presenting a disorder that compromises comprehension (e.g., dementia); pregnancy/breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility in modifying Life S-Can score | 3 months
  The outcome will be measured through the administration of Life S-Can and a quality of life questionnaire
Efficacy in improving overall quality of life | 3 months
  The outcome will be measured through the administration of Life S-Can and a quality of life questionnaire

SECONDARY OUTCOMES:
Changes in body composition | 3 months
  Changes in body composition will be measured at the end of the study by bioimpedence analysis (to detect changes in body composition). Outcome meassure will consist of weights, muscle mass, fat mass, etc.
Changes in physical activity levels | 3 months
  Changes in physical activity levels will be measured at the end of the study by administration of validated questionnaires to determine physical activity in participants. The outcome measure will be time spent doing physical activity at different levels of intensities.
Change in diet | 3 months
  Changes in diet will be measured at the end of the study by administration of validated questionnaires to determine habitual diet in participants.

OTHER OUTCOMES:
Screener validation | 3 months
  Validation of the screener (Life S-Can) will be carried out by means of administration of validated questionnaires (on physical activity, diet, alcohol intake, smoking habits, sleeping and mental health), together with objective measurements (body weight and body composition, accelerometres for physical activity, and cortisol levels in saliva).
Reproducibility of the Life S-can screener | 10 days
  Reproducibility of the screener (Life S-Can) will be measured using the retest method.
Qualitative study | The qualitative study will be carried out after the pilot intervention study and the validation of the screener have concluded. It is expected to take approximately 2 months to carry out.
  The qualitative study will determine feasibility of implementation in a clinical setting. We will evaluate and take into consideration barriers and facilitators expressed by participants to improve the implementation of the screener.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chaplin, PhD, Principal Investigator — CIBER (Consorcio Investigación Biomédica en Red); IdISBa (Fundació Instituto de Investigación Sanitaria de las Islas Baleares)
Locations (1):
- Fundació Instituto de Investigación Sanitaria de las Islas Baleares (IDISBA), Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Nogueira L, Devasia T, Mariotto AB, Yabroff KR, Jemal A, Kramer J, Siegel RL. Cancer treatment and survivorship statistics, 2022. CA Cancer J Clin. 2022 Sep;72(5):409-436. doi: 10.3322/caac.21731. Epub 2022 Jun 23. PMID 35736631
- [Background] Parry C, Kent EE, Mariotto AB, Alfano CM, Rowland JH. Cancer survivors: a booming population. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):1996-2005. doi: 10.1158/1055-9965.EPI-11-0729. PMID 21980007
- [Background] Jefford M, Howell D, Li Q, Lisy K, Maher J, Alfano CM, Rynderman M, Emery J. Improved models of care for cancer survivors. Lancet. 2022 Apr 16;399(10334):1551-1560. doi: 10.1016/S0140-6736(22)00306-3. PMID 35430022
- [Background] de Rooij BH, Park ER, Perez GK, Rabin J, Quain KM, Dizon DS, Post KE, Chinn GM, McDonough AL, Jimenez RB, van de Poll-Franse LV, Peppercorn J. Cluster Analysis Demonstrates the Need to Individualize Care for Cancer Survivors. Oncologist. 2018 Dec;23(12):1474-1481. doi: 10.1634/theoncologist.2017-0558. Epub 2018 May 8. PMID 29739897
- [Background] Dai S, Mo Y, Wang Y, Xiang B, Liao Q, Zhou M, Li X, Li Y, Xiong W, Li G, Guo C, Zeng Z. Chronic Stress Promotes Cancer Development. Front Oncol. 2020 Aug 19;10:1492. doi: 10.3389/fonc.2020.01492. eCollection 2020. PMID 32974180
- [Background] Divani A, Heidari ME, Ghavampour N, Parouhan A, Ahmadi S, Narimani Charan O, Shahsavari H. Effect of cancer treatment on sleep quality in cancer patients: A systematic review and meta-analysis of Pittsburgh Sleep Quality Index. Support Care Cancer. 2022 Jun;30(6):4687-4697. doi: 10.1007/s00520-021-06767-9. Epub 2022 Jan 26. PMID 35079904
- [Background] Alanazi MT, Alanazi NT, Alfadeel MA, Bugis BA. Sleep deprivation and quality of life among uterine cancer survivors: systematic review. Support Care Cancer. 2022 Mar;30(3):2891-2900. doi: 10.1007/s00520-021-06589-9. Epub 2021 Sep 30. PMID 34595604
- [Background] Mitchell AJ, Ferguson DW, Gill J, Paul J, Symonds P. Depression and anxiety in long-term cancer survivors compared with spouses and healthy controls: a systematic review and meta-analysis. Lancet Oncol. 2013 Jul;14(8):721-32. doi: 10.1016/S1470-2045(13)70244-4. Epub 2013 Jun 5. PMID 23759376
- [Background] Mehnert-Theuerkauf A, Hufeld JM, Esser P, Goerling U, Hermann M, Zimmermann T, Reuter H, Ernst J. Prevalence of mental disorders, psychosocial distress, and perceived need for psychosocial support in cancer patients and their relatives stratified by biopsychosocial factors: rationale, study design, and methods of a prospective multi-center observational cohort study (LUPE study). Front Psychol. 2023 Apr 20;14:1125545. doi: 10.3389/fpsyg.2023.1125545. eCollection 2023. PMID 37151329
- [Background] McDonough AL, Lei Y, Kwak AH, Haggett DE, Jimenez RB, Johnston KT, Moy B, Spring LM, Peppercorn J. Implementation of a Brief Screening Tool to Identify Needs of Breast Cancer Survivors. Clin Breast Cancer. 2021 Feb;21(1):e88-e95. doi: 10.1016/j.clbc.2020.07.006. Epub 2020 Jul 15. PMID 32807644
- [Background] Lu SC, Porter I, Valderas JM, Harrison CJ, Sidey-Gibbons C. Effectiveness of routine provision of feedback from patient-reported outcome measurements for cancer care improvement: a systematic review and meta-analysis. J Patient Rep Outcomes. 2023 Jun 5;7(1):54. doi: 10.1186/s41687-023-00578-8. PMID 37277575
- [Background] Basu A, Bhattacharya S, Miller K. A pilot study of a low-intensity health education intervention on activity and quality-of-life measures for cancer survivors. Journal of Clinical Oncology 34, no. 3_suppl (2016) 221-221.
- [Background] Cruz Bermudez, HF; Moreno Collazos, JE; Angarita Fonseca, A. Medición de la calidad de vida por el cuestionario QLQ-C30 en sujetos con diversos tipos de cáncer de la ciudad de Bucaramanga-Colombia. Enferm glob 2013 vol.12 nº30.
- [Background] Anthoine E, Moret L, Regnault A, Sebille V, Hardouin JB. Sample size used to validate a scale: a review of publications on newly-developed patient reported outcomes measures. Health Qual Life Outcomes. 2014 Dec 9;12:176. doi: 10.1186/s12955-014-0176-2. PMID 25492701
- [Derived] Chaplin A, Wordsworth J, Prohens L, Obrador-Hevia A, Guillot M, Ricci-Cabello I, Sese A, Romaguera D. Validation and pilot feasibility study of a novel screener to assess diet, lifestyle and mental health in people living with and beyond cancer: Study protocols. PLoS One. 2025 Jun 5;20(6):e0323671. doi: 10.1371/journal.pone.0323671. eCollection 2025. PMID 40472046
- See also: World Cancer Research Fund/American Institute for Cancer Research. Diet, Nutrition, Physical Activity and Cancer: a Global Perspective. Continuous Update Project Expert Report 2018. — https://www.wcrf.org/diet-activity-and-cancer/
- See also: National Comprehensive Cancer Network [Internet]. Survivorship Care for Healthy Living [cited 2023 Jul 11]. Patient resources. — https://www.nccn.org/patientresources/patient-resources
- See also: American Heart Association. Life's Essential 8. Healthy Lifestyle.2023. Accessed May16, 2023. — https://www.heart.org/en/healthy-living/healthy-lifestyle/lifes-essential-8